CLINICAL TRIAL: NCT05905744
Title: A Prospective, Multicenter Clinical Study on the Diagnostic Value of "eyeMax Insight" Cholangioscopy for Unexplained Bile Duct Stenosis
Brief Title: "eyeMax Insight" Cholangioscopy for Unexplained Bile Duct Stenosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Oriental Hepatobiliary Surgery Hospital Affiliated to Naval Military Medical University (Unknown); Zhejiang University (Other); The First Affiliated Hospital of Nanchang University (Other); West China Hospital (Other); LanZhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Peking University Cancer Hospital & Institute (Other); First Hospital of China Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Shandong Province Third hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: eyeMAX
Record Dates: First submitted 2023-05-31; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Bile Duct Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with unexplained bile duct stenosis: Patients with unexplained bile duct stenosis undergo cholangioscopy examination and ERCP
  Interventions: Diagnostic Test: cholangioscopy

INTERVENTIONS:
Diagnostic Test: cholangioscopy — cholangioscopy examination and forceps biopsy, followed by brush biopsy from ERCP

SUMMARY:
When clinical doctors cannot diagnose the cause of biliary stricture after comprehensive laboratory and imaging examinations, it is collectively referred to as unexplained bile duct stenosis. This study intends to analyze the diagnostic value of the biliary endoscopy system for unknown cause biliary strictures , and compare the diagnostic efficacy of biopsy under biliary endoscopy guidance with brushing cytology under ERCP.

DETAILED DESCRIPTION:
When clinical doctors cannot diagnose the cause of biliary stricture after comprehensive laboratory and imaging examinations, it is collectively referred to as unexplained bile duct stenosis. This study intends to analyze the diagnostic value of the biliary endoscopy system for unknown cause biliary strictures , and compare the diagnostic efficacy of biopsy under biliary endoscopy guidance with brushing cytology under ERCP.

The etiology of biliary strictures is complex, including not only malignant tumors , but also factors such as stones, inflammatory strictures, congenital variations and so on. Currently, the main methods for diagnosing malignant biliary obstruction in clinical practice include clinical examinations, biochemical testing (such as serum CA19-9), imaging, and endoscopic retrograde cholangiopancreatography (ERCP). However, these methods have limitations, such as the limited specificity and sensitivity of CA19-9 and the indirect imaging of ERCP after contrast agent filling. Therefore, these methods are relatively difficult to distinguish the benign and malignant nature of biliary lesions. This study intends to analyze the diagnostic value of the biliary endoscopy system for these unexplained bile duct stenosis.

ELIGIBILITY:
Inclusion Criteria:

Unexplained bile duct strictures (cannot be clearly diagnosed by CT, MRI or other imaging methods);

Exclusion Criteria:

* Patients with cardiac dysfunction, acute pancreatitis, active viral hepatitis;

  * Patients with mental illness; ③ Previously underwent choledochoscopy examination; ④ Malignant biliary obstruction;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with common bile duct stricture whose cause cannot be found by routine imaging and other examination methods.
Sampling Method: Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
positive rate of visual diagnosis of cholangioscopy for unexplained bile duct stenosis | 1 years
  The results are compared with pathological results of surgical specimens
positive rate of cholangioscopy-guided forceps biopsy | 1 years
  The results are compared with pathological results of surgical specimens

SECONDARY OUTCOMES:
adverse event rate of each individual technique | 1 years
  record any adverse events related to the procedure
the positive rate of biopsy | 1 years
  cholangioscopy-guided forceps biopsy, ERCP-guided brush biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Yunfeng Wang, Doctor, Principal Investigator — Changhai Hospital

IPD SHARING:
Plan to Share IPD: No